CLINICAL TRIAL: NCT01061060
Title: The Effect of Prostaglandin I2 (Beraprost Na), Administered Orally for Eight Weeks, on the Endothelial Cell Functional Disorder in Type II Diabetes Mellitus Patients With Symptoms of a Minute Peripheral Blood Flow Disorder
Brief Title: The Effect of Prostaglandin I2 on the Endothelial Cell Function Disorder in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Principal Investigator, Donghoon Choi, professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BER-CL-AKR-2009-01
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus; Peripheral Microvascular Symptoms
Keywords: Prostaglandin I2; Beraprost Na; Endothelial cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Epoprostenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beraprost group (Experimental): Prostaglandin I2
  Interventions: Drug: Prostaglandin I2
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prostaglandin I2 — oral
  Other Names: Beraprost Na
  Arms: Beraprost group
Drug: Placebo — oral
  Arms: Placebo group

SUMMARY:
This study attempts to examine the effect of oral prostaglandin I2 (Beraprost Na), administered for eight weeks, on the endothelial cell functional disorder among asymptomatic high risk diabetes mellitus patients.

DETAILED DESCRIPTION:
This study plans to include those subjects who have complaint of peripheral microvascular symptoms but have evidences of having neither a coronary arterial disease nor a peripheral arterial disease and show normal findings in the vascular stiffness test (PWV and ABI)) and plethysmography of the legs (PVR)) ,among Type II diabetes mellitus patients of forty-five (45) years old or older, This study is conducted by using a randomized double blind method. These drugs are distributed through a pharmacy in the clinical study center and administered randomly for eight weeks while this study allots patients by using a double blind method. Beraprost Na is administered along with a placebo that was manufactured by the same manufacturer to have the identical exterior look and weight of Beraprost Na. After eight weeks of drug administration, this investigation attempts to verify symptomatic improvement and change in the endothelial function by using VENDYS® and ICG perfusion imaging.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus patient
* Patients with symptoms of a minute peripheral blood flow disorder

Exclusion Criteria:

* Cases with either an already-diagnosed coronary arterial disease or a peripheral vascular disease
* Cases with a history of stroke
* Cases with an abnormal finding of vascular stiffness test (PWV and ABI) and plethysmography of legs (PVR)
* Pregnant women or fertile women with an unclear pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Symptomatic improvement by Total Symptom Score (TSS) | after 8-week treatment

SECONDARY OUTCOMES:
Change in endothelial function expressed in the unit of temperature rebound and the extent of its rise | after 8-week treatment
Change in mean rate of blood flow in the toes | after 8-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dong-Hoon Choi, Principal Investigator — Department of Internal Medicine, Severance Hospital, Yonsei Medical School, Yonsei University
Locations (1):
- Seoul, Seodaemun-gu, South Korea